CLINICAL TRIAL: NCT01144000
Title: Efficacy and Safety of Daptomycin (With or Without Rifampin) in the Treatment of Staphylococcal Hip, Knee and Shoulder Prosthetic Joint Infection
Brief Title: Daptomycin With Rifampin for Treatment of Staphylococcal Prosthetic Joint Infection
Acronym: Dapto-Studie
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Andrej Trampuz (Other)
Collaborators: University of Lausanne Hospitals (Other); Kantonsspital Liestal (Other); Schulthess Klinik (Other)
Responsible Party: Sponsor-Investigator, Andrej Trampuz, Dr. med., Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCBC134ACH03T
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Staphylococcal Infections
Keywords: Prosthetic joint infection; daptomycin; staphylococcus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daptomycin (Experimental): High dose Daptomycin in hip, knee and shoulder prosthesis infections
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — 10mg/kg/24h i.v.(intravenous) for 2-3 weeks with/or without rifampin (depending if the prosthesis is removed or not)
  Other Names: Cubicin

SUMMARY:
To determine the outcome and safety of a combined antimicrobial treatment involving daptomycin and surgical approach involving retention or short-interval two-stage exchange of the implant. Patients with hip, knee and shoulder Prosthetic Joint Infection (PJI) caused by methicillin-susceptible and methicillin-resistant staphylococci will be included and followed during 2 years.

DETAILED DESCRIPTION:
In this prospective open observational clinical study (phase 2) patients with hip, knee and shoulder PJI (as defined below) caused by methicillin-susceptible and methicillin-resistant staphylococci will be included. An informed consent will be obtained prior to patient inclusion. Medical records will be prospectively abstracted for demographic characteristics, clinical, radiographic, laboratory and microbiologic data using a standardized case report form (CRF). After inclusion, intravenous daptomycin 10 mg/kg (calculated as actual body weight) is given once daily for 2-3 weeks, followed by oral rifampin-containing antibiotics for a total of 3 months (as outlined below).

Two surgical modalities will be applied according to the PJI treatment algorithm:

* Open debridement and retention of the prosthesis (change of mobile parts): daptomycin will be combined with rifampin.
* Two-stage exchange of the prosthesis with a short interval (2-3 weeks): daptomycin of the prosthesis: daptomycin will be used alone.

The decision whether the implant will be retained or removed is based on objective criteria of the treatment algorithm and is not subject to bias. All consecutive patients with a staphylococcal PJI infection of the hip, knee or shoulder prosthesis will be included, if no exclusion criterion is present, obviating the selection bias. Since not many specialized institutions are treating patients with PJI, we expect low number of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been obtained;
2. Subject is 18-80 years of age;
3. Subject has a PJI of the hip, knee and shoulder prosthesis caused by Staphylococcus aureus or coagulase-negative staphylococci (CNS) susceptible to daptomycin and rifampin;
4. Surgical approach: Debridement and retention of the prosthesis OR a two-stage prosthesis exchange with a short interval (2-3 weeks). The selection of the surgical procedure is performed according to the PJI treatment algorithm;
5. Subject is willing to participate in the study, to follow protocol study treatment regimen, and to comply with all planned follow-up assessments;
6. Females of childbearing potential are willing to practice reliable birth control measures other than oral contraceptives (e.g., condoms or diaphragms together with a spermicidal foam or gel) and willing to undergo a urine pregnancy test prior to study entry.

Exclusion Criteria:

1. Significant renal insufficiency (creatinine clearance rate ≤30 ml/min, as determined by the Cockcroft-Gault equation at inclusion);
2. Significant hepatic dysfunction at inclusion (AST or ALT ≥4 x upper limit of normal value);
3. Elevated creatin phosphokinase (CPK) ≥2 x upper limit of normal value at inclusion
4. PJI caused by additional microorganism;
5. Non-adherence to the PJI treatment algorithm (see below);
6. Subject has been previously enrolled in the study or is currently enrolled in another investigational study previously enrolled in the study or is currently enrolled in another investigational study, which deviates from the treatment algorithm;
7. Subject had prior exposure to daptomycin within the past 3 months;
8. Allergy or intolerance to daptomycin or rifampin, known hypersensitivity;
9. Body mass index (BMI) >45 kg/m²;
10. Subject is pregnant, nursing or lactating;
11. Inability to read and understand the participant's information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy (infection-free period) | During study and 2 years after

SECONDARY OUTCOMES:
Safety of daptomycin (incidence of side effects) | During study and 2 years after
Population pharmacokinetic profile of antibiotics (daptomycin, rifampin) will be evaluated through concentration measurements in plasma and drainage fluid. | during treatment (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, Principal Investigator — Centre hospitaliere universitaire vaudvoise (CHUV) University Hospital of Lausanne
Locations (3):
- Switzerland (3):
  - Centre hospitaliere universitaire vaudois (CHUV), Lausanne, Canton of Vaud
  - Kantonsspital, Liestal
  - Schulhess Clinic, Zurich